CLINICAL TRIAL: NCT02794064
Title: Clinical Evaluation of a Prototype Tri-modal Imaging Instrument for Guiding Breast Cancer Surgery
Brief Title: A Prototype Tri-modal Imaging Device for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-8692
Record Dates: First submitted 2016-05-27; First posted 2016-06-08 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer Invasive Nos; Primary Invasive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tri-modal imaging (Experimental): Ultrasound and photoacoustic imaging of breast and adjacent lymph nodes. Imaging time: Approximately 30 minutes
  Interventions: Device: Tri-modal imaging

INTERVENTIONS:
Device: Tri-modal imaging — This tri-modal imaging system was developed in collaboration with Sogang University and is composed of three subsystems: ultrasound, photoacoustic and fluorescence. For this study, the fluorescence subsystem will not be used. The photoacoustic and ultrasound subsystems and data acquisition are controlled by a single workstation. The complete system is Canadian Standards Association (CSA) certified

SUMMARY:
Breast conservation surgery (BCS) is performed on patients with breast cancer with the intent to resect and completely remove the tumour while conserving as much of the surrounding normal tissue as possible. Currently, there is no way for surgeons to determine the adequacy of surgical resection in real-time during surgery; the assessment of surgical margins requires histological examination that is not available in real-time and is impractical in most clinical cases. This results in a re-excision rate of 23% among Canadian women in order to achieve optimal surgical margins. In addition, the presence or absence of cancer in tumor draining lymph nodes is recognized as a key element for breast cancer staging; however, lymph node dissection can be associated with overtreatment and morbidity (nerve damage and post surgical lymphedema) and histological analysis of nodes can be time consuming and thus delay subsequent procedures. In an effort to address these issues, we have designed and constructed, in collaboration with Sogang University, Seoul, S. Korea, a novel imaging system that performs three complementary imaging modalities (tri-modal): ultrasound (US), photoacoustic (PA) and fluorescence (FL).

This first-in-human pilot study will recruit 10 breast cancer patients undergoing breast conserving surgery at Princess Margaret Hospital (Toronto, Canada). The study is designed to test our tri-modal (US, PA, FL) imaging technology in breast cancer patients. The overall goal is to obtain initial information on the technical feasibility of the tri-modal system in a peri-operative setting and to confirm the anticipated safety of the procedures. Additionally, it will provide initial data on the ability of this system to detect/localize primary breast cancer lesions and cancer-involved lymph nodes prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with biopsy-confirmed first primary invasive unilateral breast cancer
* 18 years of age or older
* Have consented to standard of care surgery (lumpectomy, mastectomy) for primary invasive breast cancer, with or without auxiliary lymph node dissection
* Have had pre-surgical imaging of the affected breast and (where applicable) lymph notes (Note: additional imaging may also be done day of scheduled surgery i.e. mammography, nuclear medicine)
* Have existing biopsies banked at the hospital
* Surgery scheduled at Princess Margaret Hospital
* Tumor size of 1 cm or larger

Exclusion Criteria:

* Inability to provide informed consent
* Pre-operative therapy for current breast cancer (including chemotherapy, endocrine therapy and radiotherapy)
* history of other previous cancer requiring therapy (including chemotherapy, endocrine therapy and radiotherapy) within the past 12 months
* History of photosensitivity, skin disease or recurrent disease
* Pregnancy
* Absence of in-house biopsy in tissue bank
* Bilateral breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Detect/localize breast tumours and lymph nodes in vivo by using tri-modal imaging | Baseline (tri-modal imaging), post-surgical (pathology report); an average of 1-2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes